CLINICAL TRIAL: NCT04618536
Title: Comparison of Sun Protection Factor 30 Persistence Between Inorganic and Organic Sunscreen in Swimmer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shannaz Nadia Yusharyahya (Other)
Responsible Party: Sponsor-Investigator, Shannaz Nadia Yusharyahya, Consultant of Dermatology and Venereology, Faculty of Medicine Universitas Indonesia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-09-1037
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Sunscreen Persistence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inorganic sunscreen (Experimental)
  Interventions: Other: Organic sunscreen
- Organic sunscreen (Experimental)
  Interventions: Other: Inorganic sunscreen

INTERVENTIONS:
Other: Inorganic sunscreen — Inorganic sunscreen will be applied evenly to 2 areas on the back of the subject with a 1 cc syringe and gloved finger in an amount of 2 mg / cm2. In the first session, one area will be irradiated 20 minutes after sunscreen application. In the second session, the other area will be irradiated after the subject has swam for 1.5 hours.
  Arms: Organic sunscreen
Other: Organic sunscreen — Organic sunscreen will be applied evenly to 2 areas on the back of the subject with a 1 cc syringe and gloved finger in an amount of 2 mg / cm2. In the first session, one area will be irradiated 20 minutes after sunscreen application. In the second session, the other area will be irradiated after the subject has swam for 1.5 hours.
  Arms: Inorganic sunscreen

SUMMARY:
Prolonged sunlight exposure in swimming athletes can cause various changes in the skin; among them is sunburn. The use of sunscreen can reduce sunburn effectively. However, various types of physical activity that can trigger sweating, friction, washing with water, or sun exposure after sunscreen use can interfere with its effectiveness in the form of a decreased SPF level. The purpose of this study is to determine and compare the persistence of organic and inorganic sun protection factor 30 (SPF 30) sunscreens after 1.5 hours of swimming.

ELIGIBILITY:
Inclusion Criteria:

* Female or male swimming athletes aged 18-40 years.
* Practice swimming at least 3 times a week with a duration of 1.5-2 hours per practice in the morning or afternoon.
* Willing to be the subject of research by signing the consent.
* Do not have skin diseases.
* Do not have a history of allergies to sunscreens.

Exclusion Criteria:

* Existence of skin lesion in the test area.
* In the treatment of phototherapy.
* Using drugs with photosensitivity side effects.
* History of skin malignancy, history of photosensitivity reactions or history of disease affected by UV rays.
* Exposure to direct sunlight to the test area 24 hours before the study and during the study period.
* Absence of erythema response 24 hours after the radiation test.
* Erythema occurs in the entire test area box 24 hours after the radiation test.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
SPF change after swimming for 1.5 hours | 24 hours
  SPF of inorganic and organic sunscreen were calculated before and after swimming. The difference between SPF before and after swimming will be calculated and compared between the organic and inorganic group. SPF were calculated using minimal erythemal dose (MED) test. The test itself will be conducted in 2 days. Irradiation will be conducted on the first day and minimal erythemal dose result will be collected 24 hours after the irradiation.

SECONDARY OUTCOMES:
Inorganic sunscreen SPF | 24 hours
  SPF resulted from in vivo method, conducted before swimming. SPF were calculated using MED test. The test itself will be conducted in 2 days. Irradiation will be conducted on the first day and MED result will be collected 24 hours after the irradiation.
Organic sunscreen SPF | 24 hours
  SPF resulted from in vivo method, conducted before swimming. SPF were calculated using minimal erythemal dose test. The test itself will be conducted in 2 days. Irradiation will be conducted on the first day and minimal erythemal dose result will be collected 24 hours after the irradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Rachmani, MD, Principal Investigator — Indonesia University; Shannaz N Yusharyahya, MD, PhD, Principal Investigator — Indonesia University; Adhimukti T Sampurna, MD, Principal Investigator — Indonesia University; Respati W Ranakusuma, MD, PhD, Principal Investigator — Indonesia University; Sandra Widaty, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rachmani K, Yusharyahya SN, Sampurna A, Ranakusuma RW, Widaty S. The Comparison of Sun Protection Factor 30 Persistence Between Inorganic and Organic Sunscreen in Swimmers: Double-blind Randomized Clinical Trial. JMIR Dermatol. 2023 Jan 4;6:e41633. doi: 10.2196/41633. PMID 37632909
- [Derived] Rachmani K, Yusharyahya SN, Sampurna A, Ranakusuma RW, Widaty S. Comparison of Sun Protection Factor (SPF) 30 Persistence Between Inorganic and Organic Sunscreen in Swimmers: Protocol for a Multicenter, Randomized, Noninferiority, Split-Body, Double-Blind Clinical Trial. JMIR Res Protoc. 2022 Dec 21;11(12):e42504. doi: 10.2196/42504. PMID 36542453